CLINICAL TRIAL: NCT05111483
Title: Effects of Tupler's Technique on Postpartum Diastasis Recti and Strength Recovery of Abdominal Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/21/0509
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Diastasis Recti

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tupler's technique (Experimental): The subjects with DRA will receive Tupler's technique treatment plan for 18 weeks in which four steps will be followed.
  1. Repositioning with diastasis rehab splint :
  2. Protect the connective tissue
  3. Tupler's technique exercises (elevators, contractions, standing pelvic tilt, head lifts, leg slides, low back stretch) with 10 repetitions for each exercise.
  4. Diastasis safe exercises program to maintain the gains
  Interventions: Other: Tupler technique
- conventional therapy (Experimental): The subjects with DRA will receive conventional physical therapy treatment for 16 weeks in which researcher will follow these steps:
  1. Tie a scarf around abdomen while performing exercises
  2. Exercise program for diastasis recti abdominal muscles; sit ups, reverse sit ups, reverse trunk twist and U-seat exercises. (10 repetitions for each exercise)
  3. Respiratory rehabilitation manoeuvre
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Tupler technique — The subjects with DRA will receive Tupler's technique treatment plan for 18 weeks in which four steps will be followed.
  1. Repositioning with diastasis rehab splint :
  2. Protect the connective tissue
  3. Tupler's technique exercises (elevators, contractions, standing pelvic tilt, head lifts, leg slides, low back stretch) with 10 repetitions for each exercise.
  4. Diastasis safe exercises program to maintain the gains
  Arms: Tupler's technique
Other: conventional therapy — The subjects with DRA will receive conventional physical therapy treatment for 16 weeks in which researcher will follow these steps:
  1. Tie a scarf around abdomen while performing exercises
  2. Exercise program for diastasis recti abdominal muscles; sit ups, reverse sit ups, reverse trunk twist and U-seat exercises. (10 repetitions for each exercise)
  3. Respiratory rehabilitation manoeuvre
  Arms: conventional therapy

SUMMARY:
Diastasis rectus is the separation of the muscles along the midline of the abdomen, typically as seen in women after pregnancy. Separation is mostly larger than 2cm width at above, below or level of umbilicus. With this muscular pathology women do not feel any pain symptom just perceiving symptoms of physical discomfort, abdomen muscle weakness and its bulging. Excess weight of mother or baby and multiple birth pregnancy is the common risk factor for the DRA. Various tools will be used for the diagnosis of DRA such as vernier caliper by using centimeter ruler, diagnostic ultrasonography that give the exact measurement, pressure biofeedback unit which is used to assess the strength of weak muscles, and patient specific functional scale that used to determine the functional limitation and its improvement.

To treat the DRA conservatively, Tupler's technique and conventional physical therapy will be directed. Electrical muscular stimulations will also be given as a baseline before applying both treatments. In Tupler's technique, diastasis rehab splint and Tupler's exercises will be used whereas in conservative physical therapy, scarf tie around abdomen while performing exercises, Respiratory rehabilitation manoeuvre and abdominal muscle exercises will be used. The aim of the study is to find the the effects of Tupler's technique and conventional physical therapy treatment for abdominal muscle strength regaining and in reducing the diastasis recti among females with diastasis recti after their postpartum period. It is a Randomized clinical trial and convenient random sampling is to be used with an inclusion criterion of patients having age between 20-40 years, Both primiparous and multiparous women and Diastasis recti more than 2.5cm within 6 weeks or more postpartum. Patients will be randomly allocated into two groups, Group A will receive Tupler's technique and Group B will receive conventional physical therapy intervention. Total duration of study will be six months. Assessment will be done before and after the treatment. Pressure biofeedback unit, vernier caliper, ultrasound and patient specific functional scale are to be used to measure the outcomes. Data will be assessed by using parametric/non parametric test after completion of study.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20-40 years
* Both Primiparous and Multiparous women
* Diastasis recti more than 2.5cm within 6 weeks or more postpartum

Exclusion Criteria:

* Neurological signs, specific spinal pathology (e.g. disc lesions, malignancy, or inflammatory disease) or any other major medical pathology.
* Any complication during pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — condition happens only in females.
Enrollment: 34 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
strength of muscle | 6 months
  Pressure biofeedback is a tool designed to facilitate muscle re-education by detecting movement of the lumbar spine associated with a deep abdominal contraction in relation to an air-filled reservoir. gauge is attached increase in pressure tell more strength.
Inter-recti distance | 6 months
  through vernier caliper distance will be measured the distance between 2 arms can be checked.
Patient Specific Functional Scale | 6 months
  Patient Specific Functional Scale was developed by Stratford et al 1995 as a self-report outcome measure of function that could be used in patients with varying levels of independence. Scale is from 0 - 10.
  In Which "0" represents "unable to perform" and "10" represents "able to perform at prior level"

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michalska A, Rokita W, Wolder D, Pogorzelska J, Kaczmarczyk K. Diastasis recti abdominis - a review of treatment methods. Ginekol Pol. 2018;89(2):97-101. doi: 10.5603/GP.a2018.0016. PMID 29512814
- [Background] Thabet AA, Alshehri MA. Efficacy of deep core stability exercise program in postpartum women with diastasis recti abdominis: a randomised controlled trial. J Musculoskelet Neuronal Interact. 2019 Mar 1;19(1):62-68. PMID 30839304
- [Background] Fernandes da Mota PG, Pascoal AG, Carita AI, Bo K. Prevalence and risk factors of diastasis recti abdominis from late pregnancy to 6 months postpartum, and relationship with lumbo-pelvic pain. Man Ther. 2015 Feb;20(1):200-5. doi: 10.1016/j.math.2014.09.002. Epub 2014 Sep 19. PMID 25282439